

Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-438 10 mg Once-daily in the Treatment of Non-Erosive Gastroesophageal Reflux Disease

NCT Number: NCT02954848

Statistical analysis plan Approve Date: 09-May-2018

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.



#### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: Vonoprazan-3001

A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-438 10 mg Once-daily in the Treatment of Non-Erosive Gastroesophageal Reflux Disease

A Double-Blind, Phase 3 Study of TAK-438 (10 mg) in the Treatment of Non-Erosive Gastroesophageal Reflux Disease

#### PHASE 3

Version: Amendment2
Date: 9 May 2018

| Prepared by: |
|--------------|
| PPD |

#### Based on:

Protocol Version: Initial

Protocol Date: 31 August 2016

### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

# 1.1 Approval Signatures

Electronic signatures can be found on the last page of this document.

#### 2.0 TABLE OF CONTENTS 10 1.1 2.0 3.0 LIST OF ABBREVIATIONS......5 40 OBJECTIVES .......6 4.1 4.2 4.3 Study Design 6 5.0 5.1 5.2 5.3 6.0 DETERMINATION OF SAMPLE SIZE .......11 7.0 7 1 General Principles 12 Analysis Sets 19 7.2 7.3 7.3.1 7.3.2 Screen Failures 20 7.3.3 7.3.4 7.3.5 7.3.6 7.3.7 Analysis Sets 22 7.4 7.5 7.6 77 7.8

| 7.8.1 Primary Efficacy Endpoint(s) | 27 |
|---|---|
| 7.8.2 Secondary Efficacy Endpoint(s) | 29 |
| 7.8.3 Additional Efficacy Endpoint(s) | 30 |
| 7.9 Pharmacokinetic/Pharmacodynamic Analysis | 31 |
| 7.9.1 Pharmacokinetic Analysis | 32 |
| 7.9.2 Pharmacodynamic Analysis | 32 |
| 7.10 Other Outcomes | 32 |
| 7.11 Safety Analysis | 32 |
| 7.11.1 Adverse Events | 32 |
| 7.11.2 Clinical Laboratory Evaluations | 37 |
| 7.11.3 Vital Signs | 39 |
| 7.11.4 12-Lead ECGs | 40 |
| 7.11.5 Other Observations Related to Safety | 41 |
| 7.12 Interim Analysis | 41 |
| 7.13 Changes in the Statistical Analysis Plan | 41 |
| 8.0 REFERENCES | 42 |
| APPENDIX 1. CRITERIA FOR ELEVATED LIVER ENZYME | 43 |
| APPENDIX 2. CRITERIA FOR MARKEDLY ABNORMAL VALUES | 46 |
| LIST OF IN-TEXT TABLES | |
| Figure 4-1 Schematic of Study Design | 8 |
| Table 4-1 Schedule of Study Procedures | 9 |
| Table 7-1 Scoring for "General Health", "Physical Functioning", "Role - Physical", and " Bodily Pain" | 15 |
| Table 7-2 Scoring for "Vitality", "Social Functioning", "Mental Health", and "Role - | 1.6 |
| Emotional" | |
| Table 7-3 Coefficient for each subscale and intercept | 1/ |

#### 3.0 LIST OF ABBREVIATIONS

AE adverse event

AIDS acquired immune deficiency syndrome

ALP alkaline phosphatase
ALT alanine aminotransferase
AST aspartate aminotransferase

AUC area under the plasma concentration-time curve

BMI body mass index

C<sub>max</sub> maximum observed plasma concentration

CRO contract research organization

CYP cytochrome P450

FDA Food and Drug Administration

GCP Good Clinical Practice
GER gastroesophageal reflux

GERD gastroesophageal reflux disease
GGT gamma glutamyl transferase
HBsAg hepatitis B virus surface antigen
hCG human chorionic gonadotropin

HCV hepatitis C virus

HIV human immunodeficiency virus

H. pylori Helicobacter pylori

ICH International Conference on Harmonisation

INR international normalized ratio
IRB institutional review board
LA Classification Los Angeles Classification
LDH lactate dehydrogenase

LSBE long-segment Barrett's esophagus MAV Markedly Abnormal Values

MedDRA Medical Dictionary for Regulatory Activities
NERD non-erosive gastroesophageal reflux disease

PGx pharmacogenomics
PPI proton pump inhibitor

PT preferred term

QOL quality of life

RNA ribonucleic acid

SAE serious adverse event

SOC system organ class

SSBE short-segment Barrett's esophagus

TAK-438 vonoprazan fumarate

TEAE treatment emergent adverse event

ULN upper limit of normal

#### 4.0 OBJECTIVES

### 4.1 Primary Objectives

The primary objective of this study is to verify the superiority of TAK-438 to placebo in patients with NERD.

# 4.2 Secondary Objectives

The secondary objectives of this study are to assess the safety of TAK-438 in patients with NERD compared with that of placebo, to determine if the response after 2-week treatment with TAK-438 would allow prediction of the response after 4-week treatment with TAK-438.

### 4.3 Study Design

### <Study Design>

This is a phase 3, double-blind, placebo-controlled, parallel-group, multicenter study to verify the superiority of TAK-438 to placebo in the efficacy in patients with NERD of the modified LA Classification Grade N or M. This study consists of 1-week single-blind run-in period and 4-week double-blind treatment period. After the informed consent is obtained, placebo will be administered for 1 week in single-blind fashion as a run-in period. Upon completion of the run-in period, subject eligibility for this study will be confirmed and only subjects who meet all of the the entry criteria will be randomized in a ratio of 1:1 to receive TAK-438 10 mg or placebo for the 4-week, double-blind, treatment period.

The target number of the subjects stratified by the Central Adjudication Committee (CAC) according to endoscopic findings with the modified LA Classification Grade N or M at the start of the run-in period (Visit 1) is at least 30% (143 subjects) of the total planned number of subjects for each grade. (Enrollment of patients with either Grade N or M is to end when the number of enrolled subjects with each Grade exceeds 332 subjects, or 70% of the total planned number of subjects.)

#### <Treatment/Assessment Duration>

This study consists of a 1-week, single-blind, run-in period and a 4-week, double-blind treatment period.

#### Run-in Period

The subjects will undergo endoscopic examination within 28 days after signing of the informed consent to select patients with the modified LA Classification Grade N or M. Then, the subjects will enter the run-in period and take 1 tablet of the study drug for the run-in period (TAK-438 placebo tablet) orally once daily after breakfast for 1 week.

The study drugs to be taken during the run-in period will be prescribed after all examinations and assessments scheduled at the start of the run-in period (Visit 1) are completed. The subjects will receive the first dose of the study drug for the run-in period before leaving the sites.

#### **Treatment Period**

After subject eligibility is confirmed, the eligible subjects will be randomized to receive TAK-438 10 mg or placebo. The start date of the study drug for the treatment period is defined as Day 1.

The subjects will enter the treatment period after randomization and take 1 tablet for the treatment period (TAK-438 10 mg tablet or TAK-438 placebo tablet) orally once daily after breakfast for 4 weeks.

The study drugs to be taken during the treatment period will be prescribed after all examinations and assessments scheduled at the start of the treatment period (Visit 2) are completed. The subjects will receive the first study drug for the treatment period before leaving the sites.

After 2 weeks and 4 weeks of treatment (Visit 3 and Visit 4), the subjects are required to visit the sites without taking the study drug. After 2 weeks of treatment (Visit 3), the subjects will receive the study drug after completing all examinations and assessments scheduled for the visit, but before leaving the sites.

#### <Others>

This study will be conducted at approximately 45 sites in Japan. The planned number of subjects to be randomized is 237 per group, or 474 in total.

The subjects are required to visit the sites 4 times in total: at the start of the run-in period (Visit 1), at the start of the treatment period (Visit 2), after 2 weeks of treatment (Visit 3), and after 4 weeks of treatment (Visit 4).

Endoscopic findings will be assessed by the CAC, and the subject eligibility will be confirmed based on the decision by the investigator.

#### <Schematic of Study Design>

A schematic of the study design is included as Figure 4-1. A schedule of assessments is listed in Table 4-1.

Figure 4-1 Schematic of Study Design



<sup>\*</sup>Informed consent must be obtained within 28 days prior to the start of the run-in period (Visit 1).

**Table 4-1** Schedule of Study Procedures

| Period | Run-in Period | Т | reatment Period | | |
|---|---|---|---|---|---|
| Timing | Start of run-in period | Start of treatment period | Week 2 | Week 4 | Early termination |
| Day | Day –7 | Day 1* | Day 15 | Day 29 | _ |
| Visit Windows (Days) | −10 to −7 | 1 | 12 to 18 | 26 to 32 | Within 7 days<br>after last dose |
| Visit Number | 1 | 2 | 3 | 4 | _ |
| Informed consent (a) | X | | | | |
| Primary inclusion/exclusion criteria | X | | | | |
| Secondary inclusion/exclusion criteria | | X | | | |
| Demographics and medical history | X | | | | |
| Medication history | X | | | | |
| History of taking acid suppressants | X | | | | |
| Physical examination | X | X | X | X | X |
| Vital signs | X | X | X | X | X |
| Weight and height | X | | | | |
| Concomitant medications | <b></b> | | | | <b></b> |
| Concurrent medical conditions | X | | | | |
| Clinical laboratory tests (b) | X | X | X | X | X |
| Anti-H. pylori antibody | X (e) | | | | |
| Serum gastrin pepsinogen I/II levels | | X | X | X | X |
| PGx sample (c) | | | X (f) | | X (f) |
| Pregnancy test (hCG) (d) | X | X | X | X | X |
| ECG | X (g) | | | X | X |
| Patient diary | <b>—</b> | | | | <b>-</b> |
| QOL survey | X | X | X | X | X |
| Endoscopy | X (g) | | | | |
| Randomization | | X | | | |
| Start of study drug for the run-in period | X (h) | | | | |
| Start of study drug for the treatment period | | X (i) | | | |
| Review treatment compliance | | X | X | X | X |
| AE assessment | <b></b> | | | | <b>-</b> |

<sup>\*</sup>The start date of the study drug for the treatment period is defined as Day 1.

- (b) Hematology, chemistry, and urinalysis tests.
- (c) To be taken from subjects who gave informed consent to participate in PGx research.
- (d) To be performed only in female subjects of childbearing potential.
- (e) Anti-*H. pylori* antibody measurements need to be made between Day -10 and Day 1.
- (f) To be taken after 2 weeks of treatment as a rule, with the visit window for this sampling being from the start of the study drug in the treatment period to the end of the treatment period/the early termination of the study. In subjects who discontinue the study drug, PGx samples will be collected only in those whose samples remain to be collected at that time point.
- (g) Any results available from ECG and endoscopy performed in a routine clinical setting within 7 days prior to the start of the run-in period (before signing of informed consent) may obviate the need for ECG and endoscopy scheduled at the start of the run-in period (Visit 1).
- (h) The subject is to take the study drug for the run-in period before going home after completion of all assessments at the start of the run-in period (Visit 1).
- (i) The subject is to take the study drug for the treatment period before going home after completion of all assessments at the start of the treatment period (Visit 2).

<sup>(</sup>a) Informed consent to participate in the study will be obtained from the subjects within 28 days before the start of the run-in Period (Visit 1).

#### 5.0 ANALYSIS ENDPOINTS

### 5.1 Primary Endpoints

Heartburn during the treatment period. The following variables of the primary endpoint in the TAK-438 10 mg group are compared with those in the placebo group:

- Primary variable: proportion of days without symptoms.
- Secondary variable: cumulative rate of improvement in symptoms.
- Additional variable: severity of symptoms.

### 5.2 Secondary Endpoints

The primary endpoint is stratified as follows:

- The primary endpoint in subject subgroups stratified by the response (improved or not improved) at Week 2.
- The primary endpoint in subject subgroups stratified by endoscopic finding (Grade N or M).
- The primary endpoint in subject subgroups stratified by the combination of endoscopic finding (Grade N or M) and response (improved or not improved) at Week 2.
- The primary endpoint in subject subgroups stratified by the response (improved or not improved) to acid suppressants (proton pump inhibitors [PPIs], histamine H<sub>2</sub>-receptor antagonists [H<sub>2</sub>RAs], or other agents [anticholinergics or anti-gastrin drugs]) in subjects who had a medication history of any of these drugs.

### 5.3 Additional Endpoints

<Efficacy>

Quality of life (QOL)

Regurgitation during the treatment period

<Safety>

Treatment emergent adverse events (TEAEs), clinical laboratory test values, electrocardiogram (ECG) findings, vital signs, serum gastrin and pepsinogen I/II levels

In this study, samples for pharmacogenomics (PGx) will be collected and stored for exploratory investigation of markers enabling the prediction of drug response.

In this study using TAK-438, or in a set of clinical trials, if variability is seen in responsiveness to study drug and it is suspected to attribute its cause to subject's gene polymorphism, PGx analyses should reveal the following as required:

• Gene polymorphism and safety and/or tolerability of study drug.

Gene polymorphism and efficacy of study drug.

#### 6.0 DETERMINATION OF SAMPLE SIZE

The planned sample size is 474 subjects in total, 237 subjects for each group.

The number of evaluable subjects required for the primary endpoint will be 460 in total, 230 for each group.

### Justification of the planned sample size

In a phase 3 double-blind study of lansoprazole (AG-1749/CCT-206) evaluating the proportion of days without heartburn in those given AG-1749 15 mg and placebo, the mean proportion of days without heartburn and their standard deviations (SD) were shown to be 51.03%±28.388% in the placebo group versus 63.21%±32.200% in the AG-1749 15 mg group. Additionally, in the postmarketing study for lansoprazole (AG-1749/CCT-971), the mean proportion of days without heartburn and their SD were shown to be 46.83%±32.350% in the placebo group and 55.36%±34.545% in the AG-1749 15 mg group. In a phase 3 double-blind study of TAK-438 (TAK-438/CCT-201), the mean proportion of days without heartburn and their SD were shown to be 22.63%±28.202% in the placebo group and 28.89%±34.853% in the TAK-438 10 mg group.

Assuming that, based on these results and assessment method of heartburn in this study, the difference between the TAK-438 10 mg group and the placebo group will be 10% with a common SD of 32%, 230 subjects per treatment group will be required to ensure 90% power of the Wilcoxon rank sum test with a significance level of 5%. Thus, it is appropriate that 237 subjects will be required for each treatment group, taking into account some dropouts, 3%, after randomization.

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

### 7.1 General Principles

All statistical analyses will be conducted using

A statistical test for the primary endpoint will be reported as 1-sided and will be assessed at  $\alpha$ =0.025 significance level and all confidence intervals will be reported as 2-sided unless otherwise stated. P-values will be rounded to 4 decimal places prior to assessment of statistical significance.

Means and medians will be presented to 1 more decimal place than the recorded data. The standard deviations (SDs) will be presented to 2 more decimal places than the recorded data. Confidence intervals about a parameter estimate will be presented using the same number of decimal places as the parameter estimate.

Where appropriate, variables will be summarized descriptively by study visit. For the categorical variables, the count and proportions of each possible value will be tabulated by treatment group. The denominator for the proportion will be based on the number of subjects who provided non-missing responses to the categorical variable. For continuous variables, the number of subjects with non-missing values, mean, median, SD, minimum, and maximum values will be tabulated. Confidence intervals for continuous variables will be calculated based on t-statistics and ones for categorical variables will be based on Wald confidence intervals without using any model, unless otherwise stated.

#### 7.1.1 Study Definitions

- QTcF interval (msec): QT interval (msec) / (RR interval (sec))<sup>0.33</sup> (rounded to the nearest whole number)
- Duration of Exposure to Study Drug in Run-in Period: Date of last dose of study drug in run-in period date of first dose of study drug in run-in period + 1
- Study Drug Compliance in Run-in Period: Number of days with "Compliance of Study Drug" in diary of "Yes" during run-in period/duration of exposure to study drug in run-in period\* 100 (rounded to 1 decimal places)
- Duration of exposure to double-blind study drug (days): Date of last dose of double-blind study drug date of first dose of double-blind study drug + 1
- Double-blind study drug compliance (%): Number of days with "Compliance of Study Drug" in diary of "Yes" during treatment period/duration of exposure to double-blind study drug \* 100 (rounded to 1 decimal places)

- Assessment target period in run-in period for proportion of days without symptoms and severity of symptoms: from latest day of first dosing date in run-in period to Day -1
- Assessment target period in treatment period for proportion of days without symptoms and severity of symptoms: from Day1 to last dosing date in treatment period
- The severity in diary will be conversed as follows for analysis of severity of symptoms. No symptom = 0, No hindrance to daily activities = 1, Mild = 2, Moderate = 3, Severe = 4
- Proportion of days without symptoms: Number of days with severity of "No symptom" or "No hindrance to daily activities"/ Number of days without severity of "Not done" \* 100 (rounded to 1 decimal places)
  - In the case that the denominator is missing or 0, it will be regarded as missing.
- Severity of symptoms: (sum total of severity in diary from Day 1 to day of last dose)/
   Number of days without severity of "Not done" (rounded to 2 decimal places)
  - In the case that the denominator is missing or 0, it will be regarded as missing.
- Response to acid suppressants will be the scale as follows:
  - scale of response to PPIs, for subjects who has taken PPIs within 180 days prior to informed consent.
  - ➤ scale of response to H2RAs, for subjects who has taken H2RAs within 180 days prior to informed consent, but not PPIs.
  - > scale of response to other agents (anticholinergics or anti-gastrin drugs), for subjects who has taken only other agents (anticholinergics or anti-gastrin drugs) within 180 days prior to informed consent.
- As for response to acid suppressants, if it is "Heartburn has been resolved" or "Heartburn has
  not been resolved but relieved", we will regard it as "Improved". if it is "Heartburn has
  remained unchanged"or "Heartburn has been worsened", we will regard it as "Not
  Improved"
- The severity in QOL except "Physical Component Summary" and "Mental Component Summary" will be conversed based on Table 7-1 and Table 7-2

- The severity of "Physical Component Summary" and "Mental Component Summary" will be conversed based on following formula.
  - score = total sum of {(score for each subscale) x (coefficient for each subscale)} + intercept
  - ➤ Coefficient for each subscale and intercept is described in Table 7-3.
  - ➤ If any score in subscale is missing, score for "Physical Component Summary" and "Mental Component Summary is also missing.

Table 7-1 Scoring for "General Health", "Physical Functioning", "Role - Physical", and "Bodily Pain"

| Subscale | Severity | Score |
|----------------------|----------------------------------|-------|
| General Health | Very Poor | 26.89 |
| | Poor | 34.38 |
| | Fair | 40.40 |
| | Good | 50.27 |
| | Very Good | 58.54 |
| | Excellent | 63.38 |
| Physical Functioning | Could not do physical activities | 16.69 |
| | Quite a lot | 27.59 |
| | Somewhat | 41.45 |
| | Very little | 47.77 |
| | Not at all | 53.54 |
| Role - Physical | Could not do daily work | 21.80 |
| | Quite a lot | 27.91 |
| | Some | 40.65 |
| | A little bit | 47.42 |
| | Not at all | 54.09 |
| Bodily Pain | Very Severe | 21.68 |
| | Severe | 31.59 |
| | Moderate | 38.21 |
| | Mild | 46.10 |
| | Very mild | 52.46 |
| | None | 60.35 |

Table 7-2 Scoring for "Vitality", "Social Functioning", "Mental Health", and "Role - Emotional"

| Subscale | Severity | Score |
|--------------------|--------------------------------|-------|
| Vitality | None | 28.68 |
| | A little | 38.51 |
| | Some | 44.48 |
| | Quite a lot | 53.74 |
| | Very much | 60.01 |
| Social Functioning | Could not do social activities | 26.00 |
| | Quite a lot | 29.15 |
| | Somewhat | 37.65 |
| | Very little | 45.60 |
| | Not at all | 55.14 |
| Mental Health | Extremely | 27.59 |
| | Quite a lot | 36.30 |
| | Moderately | 44.94 |
| | Slightly | 50.72 |
| | Not at all | 56.93 |
| Role - Emotional | Could not do daily activities | 19.98 |
| | Quite a lot | 31.42 |
| | Somewhat | 42.24 |
| | Very little | 48.04 |
| | Not at all | 54.19 |

Table 7-3 Coefficient for each subscale and intercept

| Subscale and intercept | Physical Component<br>Summary | Mental Component<br>Summary |
|---|---|---|
| General Health | 0.23024 | -0.0202 |
| Physical Functioning | 0.40672 | -0.19972 |
| Role - Physical | 0.38317 | -0.16579 |
| Bodily Pain | 0.33295 | -0.15992 |
| Vitality | 0.07537 | 0.16737 |
| Social Functioning | -0.01275 | 0.27264 |
| Mental Health | -0.30469 | 0.57583 |
| Role - Emotional | -0.14083 | 0.42927 |
| intercept | 0.67371 | 4.34744 |

### 7.1.2 Definition of Study Days

When calculating Study Day relative to a reference date (ie, date of first dose of double-blind study drug [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

When calculating Follow-up Day relative to a reference date (ie, date of last dose of double-blind study drug [Follow-up Day 0]), it will be calculated as: date of observation - reference date. Hence, reference day is always Follow-up Day 0.

### 7.1.3 Definition of Study Visit Windows

All evaluable data (ie, non-missing) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used.

Clinical laboratory tests, Vital signs and, Serum gastrin pepsinogen I/II levels

| Visit Scheduled Study Day Time Interval (day | ys) |
|----------------------------------------------|-----|
|----------------------------------------------|-----|

| | (days) | Study Day | Follow-up Day |
|----------|---------------|-----------|---------------|
| Baseline | Study Day: 1 | -10 - 1 | |
| Week 2 | Study Day: 15 | 2 - 22 | < 15 |
| Week 4 | Study Day: 29 | 23 - 32 | < 15 |

# **ECG**

| <b>V</b> 7:_:4 | Scheduled Study Day Time Interval | | val (days) |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -17 - 1 | |
| Week 4 | Study Day: 29 | 2 - 32 | < 15 |

# QOL survey

| ¥7:-:4 | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Study Day | Follow-up Day |
| Start of run-in period | Study Day: -1 | -101 | |
| Start of treatment period | Study Day: 1 | 1 | |
| Week 2 | Study Day: 15 | 2 - 22 | < 15 |
| Week 4 | Study Day: 29 | 23 - 32 | < 15 |

# Weight and height and Anti-H. pylori antibody

| <b>X</b> 74 | Scheduled Study Day | Time Interval (days) | |
|-------------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -10 - 1 | |

# **Endoscopy**

| <b>X</b> 7: :, | Scheduled Study Day | Time Interval (days) | |
|----------------|---------------------|----------------------|---------------|
| Visit | (days) | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | -17 - 1 | |

### 7.1.4 Methods for Handling Missing Data

All available efficacy and safety data will be included in data listing and tabulations. No imputation of values for missing data will be performed unless otherwise specified.

• For clinical laboratory tests, values less than the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

If the year is present but the month is missing, then the month will be treated as January for the calculation.

### 7.2 Analysis Sets

The FAS, the main analysis set used for primary efficacy analysis, will be defined as all subjects who were randomized and received at least one dose of the study drug. The safety analysis set will be defined as all subjects who received at least one dose of double-blind study drug.

The per-protocol set will consist of all FAS subjects whose primary endpoint is evaluable and who had no major protocol deviation listed below:

- Subjects who did not meet inclusion criteria #3, #4, #5, #8, #9 or, #10
- Subjects who met exclusion criteria #6, #7, #8, #9, #10, #11, #12,#13, #14 or, #17
- Subjects who have violated the rules specified in section 7.3
- Subjects with double-blind study drug compliance of less than 75%
- Subjects whose emergency key was unblinded for reasons other than SUSAR
- Subjects whose duration in run-in period was 6 days or less
- Subjects whose endoscopy performance date was not satisfied with any following condition:
  - Endoscopy performed from Day -10 to -7
  - Endoscopy performed in a routine clinical setting within 7 days prior to the start of the run-in period (before signing of informed consent)

### 7.3 Disposition of Subjects

### 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form

**Analysis** 

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA version

WHO Drug version

SAS version used for creating the datasets

Analytical

Method(s): (1) Study Information

Study information shown in the analysis variables section will be

provided.

7.3.2 Screen Failures

Analysis Set: All Subjects Who Were Not Randomized

Analysis

Variable(s): Age (years)  $[Min \le -.. < 65, 65 \le -.. < 75, 75 \le -.. < -.$ 

 $\leq = Max$ 

Gender [Male, Female]

Analytical

Method(s): (1) Screen Failures

Frequency distributions for categorical variables and descriptive

statistics for continuous variables will be provided.

7.3.3 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

**Analysis** 

Variable(s): Eligibility status [Eligible for Randomization, Not

Eligible for Randomization]

Primary Reason for Subject Not [Adverse Event, Death, Lost to

Being Eligible Follow-up, Pregnancy, Protocol

Deviation, Screen Failure, Study

Terminated by Sponsor,

Withdrawal by Subject, Other]

Analytical

Method(s): (1) Eligibility for Randomization

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible,

the total number of ineligible subjects will be used as the

denominator.

### 7.3.4 Number of Subjects Randomized by Site and Treatment Group

Analysis Set: Randomized Set

Analysis

Variable(s): Randomization status [Randomized]

Stratum: Site [Site numbers will be used as

categories]

Analytical

Method(s): (1) Number of Subjects Randomized by Site and Treatment Group

Frequency distribution will be provided for each stratum by treatment

group and overall.

# 7.3.5 Disposition of Subjects

Analysis Set: Randomized Set

Analysis Double-blind study drug

Variable(s): administration status [Randomized but Not Treated]

Reason for Not Being Treated [Adverse Event, Death, Lack of

Efficacy, Lost to Follow-up, Pregnancy, Protocol Deviation, Study Terminated by Sponsor, Withdrawal by Subject, Lack of Treatment Compliance, Other]

Double-Blind Study Drug [Completed Study Drug,

Completion Status Prematurely Discontinued Study

Drug]

Reason for Discontinuation of [Adverse Event, Death, Lack of

Study Drug Efficacy, Lost to Follow-up,

Pregnancy, Protocol Deviation, Study Terminated by Sponsor, Withdrawal by Subject, Lack of Treatment Compliance, Other]

Analytical

Method(s): (1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and

CONFIDENTIAL

overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

#### 7.3.6 Protocol Deviations

Analysis Set: Randomized Set

**Analysis** 

Variable(s): Protocol Deviation [Entry Criteria, Concomitant Medication,

Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria, Major GCP

Violations]

Analytical

Method(s): (1) Protocol Deviations

Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

### 7.3.7 Analysis Sets

Analysis Set: Randomized Set

Analysis

Variable(s): Handling of Subjects and Subject [Categories are based on the

Data specifications in Handling Rules

for Analysis Data]

Analysis Sets

Full Analysis Set [Included]
Per Protocol Set [Included]
Safety Analysis Set [Included]

Analytical

Method(s): (1) Subjects Excluded from Analysis Sets

(2) Analysis Sets

Frequency distributions will be provided by treatment group for (1), and by treatment group and overall for (2). For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

## 7.4 Demographic and Other Baseline Characteristics

Analysis Set: Randomized Set

Analysis

Variable(s): Age (years)  $[Min \le -.. < 65, 65 \le -.. < 75, 75 \le -.. < -.$ 

 $\leq = Max$ 

Gender [Male, Female]

Height (cm) [Min<= - <150, 150<= - <160,

160<= - <170, 170<= - <=Max]

Weight (kg) at Baseline [Min <= - < 50, 50 <= - < 60,

60<= - <70, 70<= - <80,

 $80 \le - \le Max$ 

BMI (kg/m<sup>2</sup>) at Baseline [Min $\leq$  -  $\leq$ 18.5, 18.5 $\leq$  -  $\leq$ 25.0,

25.0<= - <=Max]

Smoking Classification [The subject has never smoked,

The subject is a current smoker,

The subject is an ex-smoker]

Consumption of Alcohol [Drink Every day, Drink a Couple

of Days Per Week, Drink a Couple of Days Per Month, Never Drink]

Consumption of Caffeine [Yes, No]

Endoscopic Finding by PI [Grade N, Grade M]

Endoscopic Finding by CAC [Grade N, Grade M, Grade A,

Grade B, Grade C, Grade D]
[Yes (Less than 3 cm) No

Barrett Mucosa [Yes (Less than 3 cm), No,

Unknown]

| Esophageal Hiatal Hernia | [Yes (2 cm or More), Yes (Less than 2 cm), No, Unknown] |
|---|---|
| Factors Which Cause Heartburn<br>and Improvement in Living Habits<br>Physical Factors | than 2 cm), 1vo, Chkhown |
| Kyphosis | [Yes, No] |
| Evident Obesity | [Yes, No] |
| Movement | |
| Forward Flexion | [Yes, No] |
| Lying in Bed | [Yes, No] |
| Other (Movement) | [Yes, No] |
| Diet | |
| Fatty Foods (Fried Foods, Stodge, etc.) | [Yes, No] |
| Carbohydrates (Grains, Potatoes, etc.) | [Yes, No] |
| Sweet Foods (Chocolate, etc.) | [Yes, No] |
| Acidic Foods (Citrus Fruits,<br>Carbonated Beverages, etc.) | [Yes, No] |
| Spices (Pepper, Curry, etc.) | [Yes, No] |
| Other (Diet) | [Yes, No] |
| Habits | |
| Smoking | [Yes, No] |
| Caffeine Ingestion | [Yes, No] |
| Drinking Alcohol | [Yes, No] |
| The above factors are not applicable, or other factors can not | [Yes, No] |
| be specified<br>Improving Lifestyle | [Yes, No] |
| Severity of Symptoms at Baseline | |
| Heartburn | [0.00, 0.00< - <=1.00, 1.00< - <=2.00, 2.00< - <=3.00, 3.00< - <=4.00] |
| Regurgitation | [0.00, 0.00< - <=1.00, 1.00< - <=2.00, 2.00< - <=3.00, 3.00< - <=4.00] |

### CONFIDENTIAL

Has subject taken PPIs within 180 [Yes, No]

days prior to informed consent?

Has subject taken H2RAs within

180 days prior to informed

consent?

Has subject taken other agents (anticholinergies or anti-gastrin drugs) within 180 days prior to

informed consent?

Response to Acid Suppressants

[Heartburn has been resolved,

Heartburn has not been resolved but relieved, Heartburn has remained unchanged, Heartburn

has been worsened]

[Yes, No]

[Yes, No]

[Improved, Not Improved]

History of *H.pylori* Eradication [Within the last year, More than

one year before, No] [Positive, Negative]

Serological Determination for

H.pylori

Gastrin (pg/mL) at Baseline Pepsinogen I/II at Baseline

[Min <= - < 200, 200 <= - < = Max]

[Min<= - <=2.0, 2.0< - <=3.0,

3.0 < - <= Max

Analytical

Method(s): (1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

# 7.5 Medical History and Concurrent Medical Conditions

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s): (1) Medical History by System Organ Class and Preferred Term

(2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided for each treatment group. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

## 7.6 Medication History and Concomitant Medications

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medication History

**Concomitant Medications** 

Analytical

Method(s): (1) Medication History by Preferred Medication Name

(2) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided for each treatment group. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

### 7.7 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Duration of Exposure to Study  $[1 \le - \le 7, 8 \le - \le Max]$ 

Drug in Run-in Period (days)

Study Drug Compliance in Run-in  $[Min \le -.. \le 50.0, 50.0 \le -.. \le 70.0,$ 

**CONFIDENTIAL** 

Period (%) 70.0<= - <90.0, 90.0<= - <=Max]

Duration of Exposure to Double- [1<= - <= 14, 15<= - <= 28,

Blind Study Drug (days) 29<= - <=Max]

Double-Blind Study Drug [Min<= - <50.0, 50.0<= - <70.0, Compliance (%) 70.0<= - <90.0, 90.0<= - <=Max]

Analytical

Method(s): (1) Study Drug Exposure and Compliance

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

### 7.8 Efficacy Analysis

### 7.8.1 Primary Efficacy Endpoint(s)

7.8.1.1 Primary Analysis

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of Days without Symptoms of Heartburn

Cumulative Rate of Improvement in Symptoms of Heartburn

Severity of Symptoms of Heartburn

Analytical

Method(s): For proportion of days without symptoms and severity of symptoms,

descriptive statistics will be used by treatment group. The point estimate of the median difference between the treatment groups will be calculated using the Hodges-Lehmann estimation. For comparisons of the treatment groups, the Wilcoxon rank sum test will be used.

For cumulative rate of improvement in symptoms, the cumulative improvement rate of symptoms during the treatment period will be calculated for each treatment group using the Kaplan-Meier method. The symptom improvement, event date and censoring date are defined below. The cumulative improvement rate in TAK-438 10 mg group will be compared to that of the placebo group using a log-rank test. Symptom improvement: symptoms experienced on less than 2 days of

the last 7 days.

Event date: the first day of confirmed symptom improvement that continued until the last day of study treatment.

Censoring date: 6 days prior to the last day with documentation of whether the subject experienced symptoms (applicable only to subjects without symptom improvement).

### 7.8.1.2 Secondary Analysis

Analysis Set: Per Protocol Set

Analysis

Variable(s): Proportion of Days without Symptoms of Heartburn

Cumulative Rate of Improvement in Symptoms of Heartburn

Severity of Symptoms of Heartburn

Analytical

Method(s): An analysis similar to the above "Primary analysis" will be performed

using the PPS to assess the robustness of the results.

#### 7.8.1.3 Adjustments for Covariates

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of Days without Symptoms of Heartburn

Cumulative Rate of Improvement in Symptoms of Heartburn

Severity of Symptoms of Heartburn

Covariate(s): Endoscopic Finding [Grade N, Grade M]

Analytical

Method(s): For proportion of days without symptoms and severity of symptoms and

severity of symptoms of heartburn, stratified wilcoxon test will applied

using endoscopic finding as covariate.

For cumulative rate of improvement in symptoms of heartburn, stratified

logrank test will applied using endoscopic finding as covariate.

#### 7.8.1.4 Examination of Subgroups

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Proportion of Days without Symptoms of Heartburn

Cumulative Rate of Improvement in Symptoms of Heartburn

Severity of Symptoms of Heartburn

Subgroup(s): Age (years)  $[Min \le -.. < 65, 65 \le -.. < 75, 75 \le -.. < -.$ 

 $\leq = Max$ 

Weight (kg) at Baseline  $[Min \le -<50, 50 \le -<60,$ 

 $60 \le -470, 70 \le -480,$ 

 $80 \le - \le Max$ 

BMI (kg/m<sup>2</sup>) at Baseline [Min $\leq$  -  $\leq$ 18.5, 18.5 $\leq$  -  $\leq$ 25.0,

 $25.0 \le - \le Max$ 

Severity of Symptoms of Heartburn [0.00, 0.00 < - <= 1.00, 1.00 < -

at Baseline <=2.00, 2.00< - <=3.00, 3.00< -

<=4.00]

Esophageal Hiatal Hernia [Yes (2 cm or More), Yes (Less

than 2 cm), No, Unknown]

Analytical

Method(s): For proportion of days without symptoms and severity of symptoms and

severity of symptoms of heartburn, descriptive statistics will be provided

for above each subgroup by treatment group.

For cumulative rate of improvement in symptoms of heartburn, the cumulative improvement rate of symptoms during the treatment period will be calculated for above each subgroup by treatment group using the

Kaplan-Meier method.

## 7.8.2 Secondary Efficacy Endpoint(s)

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of Days without Symptoms of Heartburn

Cumulative Rate of Improvement in Symptoms of Heartburn

Severity of Symptoms of Heartburn

Stratification Response at Week 2 (Criteria 1) [improved, not improved]

factor (s):

Response at Week 2 (Criteria 2) [improved, not improved]

Endoscopic Finding [Grade N, Grade M]

Endoscopic Finding and Response [Grade N and Improved, Grade N

at Week 2 (Criteria 1) and Not Improved, Grade M and

Improved, Grade M and Not

Improved]

Endoscopic Finding and Response [Grade N and Improved, Grade N

at Week 2 (Criteria 2) and Not Improved, Grade M and

Improved, Grade M and Not

Improved]

Response to Acid Suppressants [Improved, Not Improved]

Analytical

Method(s): For secondary endpoints will be performed similarly Section 7.8.1

stratified by factors except "Response to acid suppressants" on the FAS. In addition to that, same analysis will be performed stratified by factors "Response to acid suppressants" in subjects who had a medication history of any of these drugs.

When subjects are stratified by the response (improved or not improved) at Week 2, analyses will be performed on subjects stratified for both treatment groups and for the TAK-438 10 mg group only.

## 7.8.3 Additional Efficacy Endpoint(s)

7.8.3.1 QOL

Analysis Set: Full Analysis Set

Analysis

Variable(s): General Health

Physical Functioning

Role - Physical Bodily Pain

Vitality

Social Functioning

Mental Health

Role - Emotional

Physical Component Summary Mental Component Summary

Visit: Start of run-in period, Start of treatment period, Week 2, 4

Analytical

Method(s): For endpoint, summary statistics at each visit will be provided by

treatment group. Additionally, point estimate and its 2-sided 95% CI of the difference between each TAK-438 10 mg group and the placebo

group at each visit.

## 7.8.3.2 Regurgitation during the treatment period

Analysis Set: Full Analysis Set

Analysis

Variable(s): Proportion of Days without Symptoms of Regurgitation

Cumulative Rate of Improvement in Symptoms of Regurgitation

Severity of Symptoms of Regurgitation

Subgroup(s): Response at Week 2 (Criteria 1) [improved, not improved]

Response at Week 2 (Criteria 2) [improved, not improved]

Endoscopic Finding [Grade N, Grade M]

Endoscopic Finding and Response [Grade N and Improved, Grade N

at Week 2 (Criteria 1) and Not Improved, Grade M and

Improved, Grade M and Not

Improved]

**Endoscopic Finding and Response** 

at Week 2 (Criteria 2)

[Grade N and Improved, Grade N

and Not Improved, Grade M and

Improved, Grade M and Not

Improved]

Response to Acid Suppressants [improved, not improved]

Analytical

Method(s): The same analysis as described in Sections 7.8.1.1 and 7.8.2 will be

performed.

### 7.9 Pharmacokinetic/Pharmacodynamic Analysis

Not applicable

### 7.9.1 Pharmacokinetic Analysis

Not applicable

# 7.9.2 Pharmacodynamic Analysis

Not applicable

#### 7.10 Other Outcomes

Not applicable

### 7.11 Safety Analysis

#### 7.11.1 Adverse Events

### 7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Relationship to Study Drug [Related, Not Related]

Intensity [Mild, Moderate, Severe]

Analytical

Method(s): The following summaries will be provided for each treatment group.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
  - 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 4) Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
  - 5) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
  - 6) Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of


subjects)

- Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

### Number of subjects

- Summaries for 2) and 6)
  - A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.
- Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

Summaries other than 2), 3), and 6)
 A subject with multiple occurrences of TEAE will be counted only once.

### Number of events

For each summary, the total number of events will be calculated.

### 7.11.1.2 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Intensity [Mild, Moderate, Severe]

Time of Onset (day) [1<= - <=14, 15<= - <=28, 29<= -

=Max

Analytical

Method(s): The following summaries will be provided using frequency distribution

for each treatment group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term
- (9) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (10) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (11) Most Frequent Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (12) Most Frequent Non-Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

Summary tables other than (5), (6) and, (10)
 A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.
 Percentages will be based on the number of subjects in the safety

analysis set.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

• Summary table for (10)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT.

When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

- Summary table for (11)
   Most frequent TEAEs refer to PTs whose percentages are at least 2% in any one of the treatment groups.
- Summary table for (12)
   Most frequent Non-Serious TEAEs refer to PTs whose percentages are at least 5.0% in any one of the treatment groups. If no Non-Serious TEAEs exceed a frequency of 5.0%, the frequency cutoff of 2.0% will be used instead. Percentages will be based on the number of subjects in the safety analysis set.

### 7.11.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): PTE

Analytical

Method(s): The following summaries will be provided using frequency distribution.
PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 7.11.1.4 Displays of Run-in Adverse Events

Analysis Set: All Subjects Who Received Run-in Study Drug

Analysis

Variable(s): Run-in AE

Analytical The following summaries will be provided using frequency distribution.

Method(s): Run-in AEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Run-in Adverse Events by System Organ Class and Preferred Term
- (2) Drug-Related Run-in Adverse Events by System Organ Class and Preferred Term
- (3) Serious Run-in Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Number of subjects

A subject with multiple occurrences of run-in AE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of run-in AE within a PT will be counted only once in that PT.

#### 7.11.2 Clinical Laboratory Evaluations

7.11.2.1 Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Hematology

RBC WBC Hemoglobin

Hematocrit Platelets

White blood cell differentials (Neutrophils, Eosinophils, Basophils,

Monocytes, Lymphocytes)

Serum Chemistry

ALT ALP AST

GGT Bilirubin (Total Direct Bilirubin

Bilirubin)

LDH Creatine Kinase Albumin

Protein (Total Creatinine Blood Urea Nitrogen

Protein)

Uric acid Total Cholesterol Triglycerides

Glucose Potassium Sodium

Magnesium Calcium Inorganic Phosphorus

Chloride

Visit: Baseline, Week 2, 4

Analytical

Method(s): For each variable, summaries (1) to (3) will be provided by treatment group.

For applicable variables, summaries (4) and (5) will be provided by treatment group.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.


- (3) Summary of Shifts of Laboratory Test Results
  Shift tables showing the number of subjects in each category at
  baseline and each post-baseline visit will be provided.
  For each laboratory test, the laboratory values will be classified as
  "Low", "Normal" or "High" relative to the normal reference range
  provided by the central laboratory. The shift tables will be based on
  these classifications.
- (4) Number and Percentage of Subjects with Markedly Abnormal Values(MAV) of Laboratory Parameters

  Overall frequency distributions of MAV during treatment period will be provided. If a laboratory parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix 2.
- (5) Number and Percentage of Subjects with Elevated Liver Enzyme Laboratory Parameters Overall frequency distributions of elevated hepatic parameters during treatment period will be provided. Further details are given in Appendix.

#### 7.11.2.2 Urinalysis

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Protein [-, +-, 1+, 2+, 3+, 4+]

Glucose [-, 1+, 2+, 3+, 4+, 5+]

Visit: Baseline, Week 2, 4

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment group.

- (1) Number of Subjects in Categories of Urine Laboratory Test Results Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.
- (2) Summary of Shifts of Urine Laboratory Test Results


Shift tables showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

For each urine laboratory test, the laboratory values will be classified as "Normal" or " Abnormal " relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### 7.11.3 Vital Signs

7.11.3.1 Vital Signs

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Systolic Blood Pressure

Diastolic Blood Pressure

Pulse Rate

**Body Temperature** 

Visit: Baseline, Week 2, 4

Analytical

Method(s): For each variable, summaries (1) and (2) will be provided by treatment group.

For applicable variables, summary (3) will be provided by treatment group.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs Parameters

Overall frequency distributions of MAV during treatment period will be provided. If a vital sign parameter has both lower and upper

MAV criteria, analysis will be performed for each. Further details

are given in Appendix 2.

#### 7.11.4 12-Lead ECGs

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Heart Rate

RR Interval
PR Interval
QRS Interval
QT Interval
QTcF Interval

12-Lead ECG Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

Visit: Baseline, Week 4

Analytical

Method(s): For each variable other than 12-lead ECG interpretations, summaries (1)

and (2) will be provided by treatment group.

For applicable variables, summary (3) will be provided by treatment group.

For 12-lead ECG interpretation, summary (4) will be provided by treatment group.

- (1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline will be provided for each visit.
- (2) Case Plots

Plots over time for each subject will be presented.

(3) Number and Percentage of Subjects with Markedly Abnormal Values of ECG Parameters

Overall frequency distributions of MAV during treatment period will be provided. If an ECG laboratory parameter has both lower and upper MAV criteria, analysis will be performed for each. Further

details are given in Appendix 2.

(4) Summary of Shift of 12-lead ECG Interpretation Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.11.5 Other Observations Related to Safety

7.11.5.1 Serum gastrin and pepsinogen I/II levels

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Serum Gastrin

Pepsinogen I Pepsinogen II

Pepsinogen I/II Ratio

Visit: Baseline, Week 2, 4

Analytical

Method(s): For each variable, summaries (1) will be provided by treatment group.

(1) Summary of Serum gastrin and pepsinogen I/II levels and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline will be provided for each visit.

#### 7.12 Interim Analysis

Not applicable

#### 7.13 Changes in the Statistical Analysis Plan

In section 7.8.2, the description have been modified to be accordance with protocol.

# 8.0 REFERENCES

Fukuhara S, Suzukamo Y. Manual of the SF-8 Japanese version: Institute for Health Outcomes & Process Evaluation research, Kyoto, 2004

#### **Appendix 1. Criteria for Elevated Liver Enzyme**

#### **Criteria for Elevated Liver Enzyme**

All evaluable data (ie, non-missing) obtained up to Follow-up Day 14 will be used to determine whether each criteria for elevated liver enzyme in the table below is met or not. If there is more than one parameter that need to be considered for a criteria, parameter measurements taken on the same day will be used. The following abbreviations are used: LLN for lower limit of the normal range, ULN for upper limit of the normal range, ALT for alanine aminotransferase, AST for aspartate aminotransferase, Tbili for total bilirubin, and ALP for alkaline phosphatase.

| | Criteria for Eleva | ed Liver Enzyme |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| ALT > 3xULN | ALT is greater than 3 times the ULN | ALT is non-missing and less than or equal to 3 times the ULN |
| ALT > 5xULN | ALT is greater than 5 times the ULN | ALT is non-missing and less than or equal to 5 times the ULN |
| ALT > 8xULN | ALT is greater than 8 times the ULN | ALT is non-missing and less than or equal to 8 times the ULN |
| ALT > 3xULN with Tbili > 2xULN | ALT is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either ALT is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| AST > 3xULN | AST is greater than 3 times the ULN | AST is non-missing and less than or equal to 3 times the ULN |
| AST > 5xULN | AST is greater than 5 times the ULN | AST is non-missing and less than or equal to 5 times the ULN |
| AST > 8xULN | AST is greater than 8 times the ULN | AST is non-missing and less than or equal to 8 times the ULN |
| AST > 3xULN with Tbili > 2xULN | AST is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either AST is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| ALT or AST > 3xULN | Either ALT or AST is greater than 3 times the ULN | Both ALT and AST are non-missing and less than or equal to 3 times the ULN |

| | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| ALT - ACT > 5 LU N | Either ALT or AST is greater than 5 times | Both ALT and AST are non-missing and |
| ALT or AST > 5xULN | the ULN | less than or equal to 5 times the ULN |
| ALT ACT O HIN | Either ALT or AST is greater than 8 times | Both ALT and AST are non-missing and |
| ALT or AST > 8xULN | the ULN | less than or equal to 8 times the ULN |
| | | If any of the following conditions is met: |
| ALT ACT. 2 HIN | Either ALT or AST is greater than 3 times | - Both ALT and AST are non-missing and |
| ALT or AST $> 3$ xULN | the ULN and the total bilirubin is greater | less than or equal to 3 times the ULN. |
| with Tbili > 2xULN | than twice the ULN | - Total bilirubin is non-missing and less |
| | | than or equal to twice the ULN. |
| | | Either ALT is non-missing and less than or |
| ALT LACTE A LIDI | Both ALT and AST are greater than 3 | equal to 3 times the ULN, or AST is non- |
| ALT and AST > 3xULN | times the ULN | missing and less than or equal to 3 times |
| | | the ULN |
| | | Either ALT is non-missing and less than or |
| ALT LACT > F. LILN | Both ALT and AST are greater than 5 | equal to 5 times the ULN, or AST is non- |
| ALT and AST > 5xULN | times the ULN | missing and less than or equal to 5 times |
| | | the ULN |
| | | Either ALT is non-missing and less than or |
| ALT and AST > 8xULN | Both ALT and AST are greater than 8 | equal to 8 times the ULN, or AST is non- |
| ALI and ASI > 8XULN | times the ULN | missing and less than or equal to 8 times |
| | | the ULN |
| | | If any of the following conditions is met: |
| | | - ALT is non-missing and less than or |
| ALT and AST > 3xULN with Tbili > 2xULN | Both ALT and AST are greater than 3 | equal to 3 times the ULN |
| | times the ULN and the total bilirubin is | - AST is non-missing and less than or |
| | greater than twice the ULN | equal to 3 times the ULN |
| | | - Total bilirubin is non-missing and less |
| | | than or equal to twice the ULN |
| ALD > 2III N | ALD is greater than 2 times the LH N | ALP is non-missing and less than or equal |
| ALP > 3xULN | ALP is greater than 3 times the ULN | to 3 times the ULN |

| | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| | | Either ALP is non-missing and less than or |
| ALP > 3xULN | Both ALP and ALT are greater than 3 time | equal to 3 times the ULN, or ALT is non- |
| with ALT > 3xULN | the ULN | missing and less than or equal to 3 times |
| | | the ULN |
| | | Either ALP is non-missing and less than or |
| ALP > 3xULN | Both ALP and AST are greater than 3 | equal to 3 times the ULN, or AST is non- |
| with AST > 3xULN | times the ULN | missing and less than or equal to 3 times |
| | | the ULN |

#### Classifying Subjects for the Overall Treatment Period

For each criteria and subject, classifications will be made according to the conditions i) to iii) provided below.

- i) A subject who met criteria (a) at least once after baseline will be considered to have met the criteria for elevated liver enzyme.
- ii) If condition i) is not met but if criteria (b) is met at least once after baseline, then the subject will be considered to have not met the criteria for elevated liver enzyme.
- iii) If neither i) nor ii) is met, then the subject will be excluded from the analysis for the criteria for elevated liver enzyme.

### **Appendix 2. Criteria for Markedly Abnormal Values**

# Hematology, Serum Chemistry, Vital Signs, and 12-lead ECG (except Upper MAV Criteria of QTcF Interval)

For each parameter, all evaluable data obtained up to Follow-up Day 14 will be classified as a MAV or not. The criteria in the table below will be used. The lower limit of the normal range and the upper limit of the normal range are abbreviated as LLN and ULN.

# <u>Hematology</u>

| D | Gender | Age | MAV Criteria | |
|---|---|---|---|---|
| Parameter | | | Lower Criteria | Upper Criteria |
| RBC ( $\times 10^6/\mu$ L) | - | - | <0.8×LLN | >1.2×ULN |
| Platelets ( $\times 10^3/\mu L$ ) | - | - | <75 | >600 |
| WBC ( $\times 10^3/\mu$ L) | - | - | <0.5×LLN | >1.5×ULN |
| Neutrophils (%) | - | - | <0.5×LLN | >1.5×ULN |
| Eosinophils (%) | - | - | - | >2×ULN |
| Basophils (%) | - | - | - | >3×ULN |
| Lymphocytes (%) | - | - | <0.5×LLN | >1.5×ULN |
| Monocytes (%) | - | - | - | >2×ULN |
| Hematocrit (%) | | | <0.8×LLN | >1.2×ULN |
| Hemoglobin (g/dL) | | | <0.8×LLN | >1.2×ULN |

# Serum Chemistry

| n . | Gender | Age | MAV Criteria | |
|-----------------------------|--------|-----|----------------|----------------|
| Parameter | | | Lower Criteria | Upper Criteria |
| Total protein (g/dL) | - | 1 | <0.8×LLN | >1.2×ULN |
| Albumin (g/dL) | - | ı | <2.5 | - |
| Blood urea nitrogen (mg/dL) | - | ı | - | >30 |
| Urate (mg/dL) | - | ı | - | >13.0 |
| Creatinine (mg/dL) | - | ı | - | >2.0 |
| Total cholesterol (mg/dL) | - | ı | - | >300 |
| Triglycerides (mg/dL) | - | ı | - | >2.5×ULN |
| Total bilirubin (mg/dL) | - | - | - | >2.0 |

| D | Gender | Age | MAV Criteria | |
|---|---|---|---|---|
| Parameter | | | Lower Criteria | Upper Criteria |
| Sodium (mEq/L) | - | - | <130 | >150 |
| Potassium (mEq/L) | - | - | <3.0 | >6.0 |
| Chloride (mEq/L) | - | - | <75 | >126 |
| Calcium (mg/dL) | - | - | <7.0 | >11.5 |
| Inorganic phosphorus (mg/dL) | - | - | <1.6 | >6.2 |
| Alkaline phosphatase (U/L) | - | - | - | >3×ULN |
| Creatine kinase (U/L) | - | - | - | >5×ULN |
| AST (U/L) | - | - | - | >3×ULN |
| ALT (U/L) | - | - | - | >3×ULN |
| GGT (U/L) | - | - | - | >3×ULN |
| Glucose (mg/dL) | - | - | <50 | >350 |
| Magnesium (mg/dL) | - | - | <1.2 | >3.0 |
| Direct bilirubin (mg/dL) | | | | >2×ULN |

# Vital Signs

| D | Gender | Age | MAV Criteria | |
|---|---|---|---|---|
| Parameter | | | Lower Criteria | Upper Criteria |
| Systolic Blood Pressure (mmHg) | - | ı | <85 | >180 |
| Diastolic Blood Pressure (mmHg) | - | - | < 50 | >110 |
| Pulse Rate (bpm) | - | - | < 50 | >120 |
| Body temperature (°C) | - | - | <35.6 | >37.7 |

# 12-lead ECGs

| D | Gender | Age | MAV Criteria | |
|----------------------|--------|-----|----------------|----------------|
| Parameter | | | Lower Criteria | Upper Criteria |
| Heart Rate (bpm) | - | - | < 50 | >120 |
| QT Interval (msec) | - | - | <=50 | >=460 |
| QTcF Interval (msec) | - | - | <=50 | - |

#### **Classifying Subjects for the Overall Treatment Period**

For each parameter and subject, classifications will be made according to the conditions i) to iii) provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

#### 12-lead ECG (Upper MAV Criteria of QTcF Interval)

All evaluable data obtained up to Follow-up Day 14 will be classified as a MAV or not. The criteria in the table below will be used. Note that the observed value and the change from baseline used for classification should be measurements taken on the same day.

For each subject, classifications will be made according to the conditions i) to iii) provided below.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that meets any of the following will be considered as a subject without MAV.
  - Observed value is less than 450 msec and not missing.
  - Change from baseline is less than 30 msec and not missing, and observed value is less than 500 msec and not missing.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV.

| Doromator | MAV Criteria | |
|---|---|---|
| Parameter | Lower Criteria | Upper Criteria |
| | | If either of the following conditions is met: |
| QTcF Interval (msec) | ıl (msec) | • observed value >=500 |
| | | • change from baseline >= 30 and observed value >=450 |